CLINICAL TRIAL: NCT00717990
Title: A Phase II Study of Irinotecan, Capecitabine and Avastin in Patients With Metastatic Colorectal Cancer, Who Have Progressed After 1ST Line Therapy With Folfox/Avastin.
Brief Title: Irinotecan, Capecitabine and Avastin for Metastatic Colorectal Cancer as Salvage Treatment
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor Accrual
Sponsor: University Hospital of Crete (Other)
Responsible Party: Principal Investigator, Vassilis Georgoulias, MD, MD, University Hospital of Crete
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT/05.35
Record Dates: First submitted 2008-07-16; First posted 2008-07-18 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Colorectal cancer; Bevacizumab; XELIRI
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine; Bevacizumab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): XELIRI/Avastin
  Interventions: Drug: Capecitabine; Drug: Bevacizumab; Drug: Irinotecan

INTERVENTIONS:
Drug: Capecitabine — Capecitabine 2000 mg/m2 p.o. daily, for days 1-14, every 3 weeks for 6 cycles
  Other Names: Xeloda
Drug: Bevacizumab — Bevacizumab 7.5 mg/kg intravenous (IV) on day 1 every 3 weeks for 6 cycles
  Other Names: Avastin
Drug: Irinotecan — Irinotecan 250 mg/m2 IV on day 1 every 3 weeks for 6 cycles
  Other Names: Campto; CPT-11

SUMMARY:
This study will evaluate the efficacy of Irinotecan,Capecitabine and Avastin combination in patients with no response to previous treatment with 5-Fluorouracil,Leucovorin,Eloxatin and Avastin.

DETAILED DESCRIPTION:
The aim of this phase II study is to evaluate the efficacy of the combination XELIRI/AVASTIN in patients with mCRC, who have progressed in first line treatment with FOLFOX/AVASTIN. For AVASTIN was selected the dosing schedule of the trials TREE 1 and 2 [17], where Avastin was combined with capecitabine and oxaliplatin in a three weeks schedule and with adaptation of the dose in the 7,5 mg/kg

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed locally advanced or metastatic colorectal cancer
* Measurable or evaluable disease according to the Response Evaluation Criteria in Solid Tumors
* ECOG performance status ≤ 2
* Age 18 - 72 years
* Patients who progress after 1st line therapy with FOLFOX/AVASTIN
* Adequate liver (Bilirubin ≤ 1.5 upper normal limit, SGOT/SGPT ≤ 4 upper normal limit, ALP ≤ 2.5 upper normal limit) renal (Creatinine ≤ 1.5 upper normal limit) and bone marrow (ANC ≥ 1,500/mm3, PLT ≥100,000/mm3) function
* Patients must be able to understand the nature of this study
* Written informed consent

Exclusion Criteria:

* History of serious cardiac disease (unstable angina, congestive heart failure,uncontrolled cardiac arrhythmias)
* History of myocardial infarction or stroke within 6 months
* Clinically significant peripheral vascular disease
* History of abdominal fistula, gastrointestinal perforation or intraabdominal abscess within 28 days prior to Day 0
* Major surgical procedure, open biopsy, or significant traumatic injury within 30 days prior to Day 1
* Presence of central nervous system or brain metastasis
* Evidence of bleeding diathesis or coagulopathy
* Blood pressure > 150/100 mmHg
* Pregnant or lactating woman
* Life expectancy < 3 months
* Previous radiotherapy within the last 4 weeks or > 25% of bone marrow
* Metastatic infiltration of the liver > 50%
* Patients with chronic diarrhea (at least for 3 months) or partial bowel obstruction or total colectomy
* Active infection requiring antibiotics on Day 1
* Second primary malignancy, except for non-melanoma skin cancer and in situ cervical cancer
* Psychiatric illness or social situation that would preclude study compliance

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | up to 6 months

SECONDARY OUTCOMES:
Time To Progression | 1 year
Toxicity profile | Toxicity assessment on each chemotherapy
Quality of life | Assessment every two cycles
Symptoms improvement | Assessment every two cycles
Overall Survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Vassilis Georgoulias, MD, Principal Investigator — University Hospital of Crete, Dep of Medical Oncology
Locations (1):
- University Hospital of Crete, Dep of Medical Oncology, Heraklion, Greece